







Version 2.0 20-Feb-19

Name of Person taking consent

Centre:

REC Number:

IRAS ID: 256260

## PARTICIPANT CONSENT FORM

PIN:

## This consent form is for young people aged 16+

## Online PTSD treatment for Young People and their Carers (OPTYC): Case Series Dr Patrick Smith

| | | | Please initial box |
|---|---|---|---|
| 1. | I confirm that I have read the information sheet dated 20/02/18 (version 2.0) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | |
| 3. | I understand that relevant data collected during the study may be looked at by individuals from King's College London, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | | |
| 5. | I understand that my relevant confidential information will be disclosed to appropriate professionals, including my GP, if a clinical or research worker on the study becomes concerned about my own, or someone else's safety. | | |
| 6. | I agree to my General Practitioner being informed of my participation in the study and being involved in the study, including any necessary exchange of information about me between my GP and the research team. | | |
| 7. | I understand that the information held and maintained by South London and Maudsley NHS Foundation Trust may be used to help contact me or provide information about my health status. | | |
| 8. | s. I agree to take part in the above study. | | |
| lam | e of Participant | Date | Signature |

Date

Signature